CLINICAL TRIAL: NCT04858555
Title: Staging System in Amyotrophic Lateral Sclerosis
Acronym: Biostaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I16017_1 (Biostaging)
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; ALS; Staging; Biomarker
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be collected from ALS incident cases. Neurofilaments levels will be determined in the plasma using ELISA Method
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Recently two staging systems have been proposed for amyotrophic lateral sclerosis (ALS), based on clinical milestones The King's college clinical staging system (1) and ALS Milano-Torino Staging (ALS-MITOS) (2). Further research to validate and develop an accurate staging system in different populations will improve our understanding of its pathogenesis, disease activity and progression.

General objective : To validate the two previously proposed staging system and to test the interest of considering Neurofilament biomarkers in these systems.

Specific objectives: 1) To validate the two classification systems in an independent cohort of patients with ALS followed-up in the ALS expert center of Limoges (France) 2) To assess the interest of Nf biomarkers to predict neurological decline

DETAILED DESCRIPTION:
Amyotrophic lateral sclerosis (ALS) is a rare, fatal neurodegenerative disease of the human motor system. Recently two new staging systems have been proposed for ALS, based on clinical milestones related also to the spreading pattern of the disease (1,2). Furthermore, biomarker development is still an essential component of future therapeutic development in ALS. Thus, it is also important to acknowledge the value of biomarker research in supporting or revealing fundamental pathophysiological mechanisms in ALS.

The proposed staging systems: have been recently tested in two independent cohorts (3,4) with results that were not fully consistent (ii) did not considered the potential value of biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* ALS cases recruited for retrospectively (between) 2007 to 2016 for the retrospective cohort
* ALS cases recruited for prospectively by the ALS expert center of Limoges for one year.

Exclusion Criteria:

* Previous neurosurgical operations
* A recent history of neurotrauma
* Peripheral neuropathies
* ALS/frontotemporal dementia (ALS/FTD)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients with ALS, followed-up in the ALS expert center of Limoges university Hospital (France).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-12-02 (Estimated); Study Completion 2024-12-02 (Estimated)

PRIMARY OUTCOMES:
To validate the two previously proposed staging system and to develop an accurate staging system in ALS considering Neurofilament (Nf) biomarkers. | 2 years
  To validate the two previously proposed staging system and to develop an accurate staging system in ALS considering Neurofilament (Nf) biomarkers

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Limoges University Hospital, Limoges
  - Tours University Hospital, Tours